CLINICAL TRIAL: NCT04413682
Title: Effectiveness of Structured Exercise Program on Quality of Life and Activities of Daily Living in Persons With Multiple Sclerosis: Telerehabilitation vs Supervised Program
Brief Title: Telerehabilitation vs Supervised Exercises in MS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Collaborators: Istanbul University - Cerrahpasa (Other); Medipol University (Other)
Responsible Party: Principal Investigator, Ela Tarakci, Professor, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MS-TeleRehab2019
Record Dates: First submitted 2020-05-30; First posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-05

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Telerehabilitation; Supervised exercises; Structured exercise; Quality of Life; Activities of Daily Living
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will randomly assign to the structured supervised exercise or structured home-based groups. Randomization are done using Microsoft Excel 'RAND()' function.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supervised Exercise Group (Experimental): One session per day, 3 days per week over a 12-weeks structured exercise program under supervision of a physical therapist.
  Interventions: Behavioral: Structured Supervised Exercise
- Telerehabilitation Group (Experimental): One session per day, 3 days per week over a 12-weeks structured exercise program through Telerehabilitation
  Interventions: Behavioral: Structured telerehabilitation

INTERVENTIONS:
Behavioral: Structured Supervised Exercise — Structured Exercise Program under the supervision of Physical Therapist
  Arms: Supervised Exercise Group
Behavioral: Structured telerehabilitation — Structured Exercise Program checked and controlled through telerehabilitation
  Arms: Telerehabilitation Group

SUMMARY:
Multiple sclerosis (MS) is a complex neurodegenerative autoimmune disease. People with MS (PwMS) have low quality of life (QoL) and activities of daily living (ADL). Exercise is a safe and effective rehabilitation tool for PwMS. A structured and personalized exercise program can improve physical fitness, functional capacity, quality of life and modifiable disorders in PwMS. On the other hand, Telerehabilitation is an alternative rehabilitation method in PwMS. The purpose of this study is to investigate the effectiveness of exercise programs and telerehabilitation on ADL and QoL in PwMS, and compare the effects of supervised exercise and home-based exercise programs for the PwMS.

DETAILED DESCRIPTION:
Participants are randomly assigned to the structured supervised exercise or structured home-based groups. Interventions in Group 1 (n=15) includes one session per day, 3 days a week over a 12-weeks structured exercise program under the supervision of a physical therapist. Group 2 (n=15) includes a 12-week structured home-based exercise program checked and controlled through telerehabilitation three times a week. All measurements pre-post intervention.

ELIGIBILITY:
Inclusion Criteria:

patients with:

1. Stable period at the time of application to the clinic
2. Expanded Disability Status Scale Levels between 2 - 6.5
3. Appropriate cognitive level to understand the exercises
4. No diseases to affect their participation in exercise programs

Exclusion Criteria:

patients with:

1. Poorly controlled diabetes, hypertension or other medical conditions to be incompatible with study participation,
2. A new history of previous attacks
3. No reliable informed consent

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-02-10 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
Functional Independence Measure (FIM) | Changes after 12 weeks
  FIM is a tool used for evaluation of primary ADL of people with disability. FIM items include self care, sphincter control, transfers, locomotion, communication, and social cognition subgroups. Grading is based on 7 points. 7: complete independence, 6: modified independence, 5, 4 and 3: modified dependence, 2 and 1: complete dependence.
Nottingham Health Profile, First section (NHP-I) | Changes after 12 weeks
  NHP is a tool used for measuring and definition of QoL regarding the health status in general. NHP-I contains 38 yes/no statements, focusing on different aspects of the general health problems, including six dimensions of subjective health defined as physical abilities, pain, sleep, energy, emotional reaction, energy level and social isolation. Questions are evaluated according to the patients' yes/no responses and are scored between 0 and 100. High scores indicate high level health status in the specified item. Total scores are summed in all fields.
Quality of life scale (QoLS) | Changes after 12 weeks
  QoLS is a standardized interview consisting of 41 questions clustered in four subscales: functional and economic scale, social and recreational scale, affect and life in general scale, and medical problems scale. Each question in the scale is evaluated over 5 points. (1 is negative at all times and 5 is the best response).

CONTACTS AND LOCATIONS:
Overall Officials: Ela Tarakci, Professor, Principal Investigator — etarakci@istanbul.edu.tr
Locations (1):
- Istanbul University-Cerrahpaşa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No